| | IRB Approved: 03/13/201<br>IRB Accepted: 04/10/201 | |
|---|---|---|
| Lifespan Affiliate Site where r | esearch will be conduct | ted |
| ⊠ Rhode Islan ☐ Bradley Ho | | ☐ The Miriam Hospital ☐ Newport Hospital ☐ Gateway Healthcare |

# Agreement to Participate in a Research Study And Authorization for Use and Disclosure of Information

| 005418 | |
|-------------|-------------------------|
| Committee # | Name of Study volunteer |

# **Working Memory in Overweight Children**

You and your child are being asked to take part in a research study. All research studies at Lifespan hospitals follow the rules of the state of Rhode Island, the United States government and Lifespan. Before you decide whether to participate and to allow your child to be in the study, you and the researcher will engage in the "informed consent" process. During this process, the researcher will explain the purpose of the study, how it will be carried out, and what you and your child will be expected to do if you participate. The researcher will also explain the possible risks and benefits of being in the study, and will provide other information. You should feel free to ask any questions you might have. The purpose of these discussions is for you to decide whether participating in the study is the best decision for you and your child.

If you decide to participate and to allow your child to be in the study, you will be asked to sign an agreement which states that the study has been explained, that your questions have been answered, and that you agree to participate and to have your child participate. You will be given a copy of this form to keep.

Federal and Lifespan institution rules require that if your child is 8 years or older, the "assent" (agreement) of your child be obtained by the researcher before your child may participate in this study. Your child must sign the consent form as well. You will be given a copy of the signed consent form to keep.

#### 1. Nature and Purpose of the Study

You and your child is being asked to take part in a research project because we are interested in understanding more about brain functioning and working memory in overweight children, and how this may relate to their eating behaviors. We want to better understand this process so we can help children develop better skills in these areas to improve their eating behaviors.

We expect to enroll 30 children and a parent into this study. The study is sponsored by the Rhode Island Neuroscience Leadership Committee and the Weight Control and Diabetes Research Center.

# 2. <u>Explanation of Procedures</u>

Participation will involve a screening conversation via telephone and mail to determine study eligibility. You have already completed this screening. If you and your child are eligible, you are now being asked to sign this consent form. This consent form and assent form for children will be explained to you by a member of the research team. Should you wish to participate and to allow your child to participate, you and your child will be asked to sign this consent document. You and your child will also be asked to complete several questionnaires that will determine if they are eligible for this study.

If your child is eligible and you both have agreed to participate, you and your child will be asked to stay at the Weight Control and Diabetes Research Center for approximately 2 hours for an assessment visit. During this time, you and your child will have height and weight measured, and you and your child will complete several questionnaires, interviews, and tasks about his or her eating habits and psychological functioning. We will collect information about you for the purposes of this research. This includes your name, your address, phone number, e-mail address, gender, and your child's age and date of birth.

We would like to record the interviews for training purposes, but you can decline to have them recorded.

# I GIVE THE RESEARCHERS PERMISSION TO AUDIO/VIDEORECORD THE INTERVIEWS WITH MY CHILD

| □ YES | $\square$ NO | | |
|-------------------------------|--------------|-----|------------------|
| Signature of parent/guardian* | Date | and | Time when signed |
| Signature of parent/guardian* | | and | Time when signed |

You will be given the opportunity to review the questionnaires before they are administered to your child, and to withdraw your consent for your child to complete any or all of the questionnaires if you choose. In addition, you and/or your child will be asked to complete a questionnaire which addresses how physically developed your child has become, in terms of genital (penis, testicle, or labial) growth, the emergence and growth of hair around the genitals and under the arms, as well as other parts of the body, and the appearance of breasts in girls. This is called Tanner staging, allowing the doctor and the researchers to understand at what point in physical growth towards an adult body a child or adolescent has reached.

After the assessment visit, your child will then come back for a second 2-hour visit to participate in a MRI scan at Brown University while they are viewing different words and responding during a task designed to assess their memory. An MRI scanner uses a magnet and radio waves to take pictures of your child's brain. Your child will need to lie still for the scanner for up to an hour. Being in the MRI scanner will not be painful for your child, but some

children get antsy or nervous being in the scanner, and some children become anxious or claustrophobic from lying in an enclosed space. Someone will be in a room close by while they are in the scanner, and your child will be able to tell them if s/he wants to come out. Your child will have to remove any metal items they are wearing or have on, like jewelry, cell phones, or coins. They also need to make sure they don't wear any clothes with metal zips, fasteners, buttons, belts or buckles. Make sure to tell someone if your child has an artificial limb or joint, a pacemaker, or screws or plates in their body from a previous surgery. This is because the magnet in the MRI scanner is very strong so if it comes in contact with any metal it could be dangerous for your child. You will be asked to complete an additional consent form which describes the risks and benefits of MRI procedures in greater detail.

We think you will be in the study for about 2-3 weeks, starting from the time we spoke to you on the phone, until you finish the two in-person study visits. The two visits will take about 2 hours each. We will try to schedule your visits close together so it's easier for you.

Your child will receive \$75 in cash at the end of each study visit for participating in this study (\$150 total).

<u>Costs for participating in this study</u>: There will be no costs to you or your insurance company resulting from your participation in this research study. However, you or your insurance company will be responsible for costs related to your usual medical care.

#### Contact Information:

Andrea Goldschmidt, PhD (401-793-8251; 196 Richmond St., Providence, RI, 02903) will be available to answer questions for research study volunteers about the study or any concerns about side effects /problems.

#### 3. Discomforts and Risks

Some of the questions from the interviews and questionnaires may be upsetting to you or your child. You can refuse to answer any questions you wish, ask to have the evaluation stopped at any time, or contact the investigator or research staff at (401) 793-8283 for further assistance.

This study is neither designed nor intended to detect health problems in your child. The MRI scans that your child will undergo do not substitute for an appropriate medical examination by a qualified health care provider. If you suspect that your child might be suffering from injury or illness, including any injury involving the head or brain, you should not rely on this study as a way to determine whether or not your child is well.

The investigators for this project are not trained to perform radiological diagnosis, and the MRI scans performed in this study are not designed to find abnormalities. The investigators and Brown University are not responsible for failure to find existing abnormalities in your child MRI scans. However, on occasion the investigator may notice an MRI image that seems abnormal. When this occurs, the investigator will inform you and recommend that you consult with your child's primary care physician. The decision whether to proceed with further examination or treatment lies solely with you and your physician. The investigators

and Brown University are not responsible for any examination or treatment that you undertake based upon these findings.

Because the images collected in this study do not comprise a proper clinical MRI study, these images will not be made available for diagnostic purposes.

Other possible risks include the remote possibility that the information would be released outside of the research setting, which could be upsetting for you. However, strong measures are taken to ensure that all information remains confidential. Specifically, all participants will be identified only by code number which will appear on documents used for evaluation for statistical analyses. All records and information will be kept locked in the clinical research facilities. Publications of this research will not identify individual participants.

If any mental health related problem is detected, such as suicidality, intent to harm others, or drug abuse, or if previously unreported abuse is discovered, you and/or your child will be further evaluated and steps will be taken to ensure their safety (e.g., creating a safety plan, providing referrals). Reports of physical or sexual abuse will be reported to state authorities as mandated by law.

There may be other risks that could arise which are not reasonably foreseeable. If new information becomes available which could influence your willingness to continue, this new information will be discussed with you.

#### 4. Benefits

If you and your child agree to take part in this study, there may or may not be direct benefit to you and your child. We hope the information learned from this study may benefit overweight children in the future or aid in our understanding of working memory in overweight children.

# 5. Alternative Therapies

Since treatment is not being offered, there are no alternative therapies. You may choose not to participate. The decision whether or not you wish to participate in this study will not affect your care at Lifespan.

### **6.** Refusal/Withdrawal

It is up to you whether you want your child to be in the study. You are not required to enroll your child or participate. If you decide you want your child to participate, you can always change your mind and remove them from the study at any time. If you decide not to have your child be in the study, or if you remove them later, your child will still be able to get the health care services they would normally get. If you enroll your child but later on the researcher or your doctor feels being in the study is no longer good for your child, they may choose to take your child out of the study before it is over. If new information becomes available that might change your mind about whether you want your child to stay in the study the researcher will share this information with you as soon as possible.

Taking part in this study is voluntary. If you choose not to participate in this study, your care at Lifespan will not be affected.

You may choose not to participate at any time during the study. Leaving the study will not affect your care at Lifespan.

If you choose to no longer be in the study and you do not want any of your future health information to be used, you must inform Dr. Goldschmidt in writing at the address on the first page. Dr. Goldschmidt may still use your information that was collected prior to your written notice.

Dr. Goldschmidt may decide to take you out of the study without your consent if:

- Your child is unable to meet the requirements of the study;
- Your child's medical condition changes;
- New information becomes available that indicates that participation in this study is not in your child's best interest; or
- If the study is stopped, or the sponsor chooses to end the study. This may happen at any time, for reasons unrelated to healthcare.

## 7. Medical Treatment/Payment in Case of Injury

A research injury is any physical or mental injury or illness caused by being in the study. If your child is injured by a medical treatment or procedure they would have received even if they were not in the study that is not a research injury. To help avoid research injury and added medical expenses, it is very important to follow all study directions carefully. If your child does experience a research injury, Lifespan or the study doctor can arrange medical treatment for them. Such treatment will be paid for as described below.

If you suffer an unanticipated injury as a direct result of this research and require emergency medical treatment, Lifespan will provide such treatment at no cost to you. You must notify Dr. Goldschmidt as promptly as possible after your injury in order to receive this care. An injury is "unanticipated" if it is not one of the known effects of a study drug, medical device or procedure, and is not the result of your disease or condition. The costs of any non-emergency care for such an injury will be billed to you or your insurance in the ordinary manner. If you think that you have suffered a research related injury, you must let Dr. Goldschmidt know right away.

If you have insurance and your child has a research injury that is not covered by the study, it is possible that some or all of the cost of treating your child could be billed to your insurer. If your health insurance will not cover such costs, it is possible you would have to pay out of pocket. In some cases, Lifespan might be able to help you pay if you qualify for free care under Lifespan policy. However, Lifespan has no policy to cover payment for such things as lost wages, expenses other than medical care, or pain and suffering.

#### **8.** Rights and Complaints

Signing this form does not take away any of your lawful rights. If you or your child have any complaints about your child's participation in this study, or would like more facts about the rules for research studies, or the rights of people who take part in those studies, you may contact Janice

Muratori, anonymously if you wish, in the Lifespan Office of Research Administration, telephone number (401) 444-6246.

# 9. <u>Confidentiality and Research Authorization for Use and Disclosure of Your Health Care</u> Information.

Your child's research records will be treated as private health care records and will be protected according to Lifespan privacy practices and policies that are based on state and federal law. In particular, federal law requires us to get your permission to use or disclose (release your child's information to someone outside of Lifespan) their health information for research purposes. If you sign this form you agree to have your child be in this research study and you permit the use and disclosure of your child's health information for the purpose of conducting the research, providing treatment, collecting payment and running the business of the hospital. This permission has no expiration date. You may withdraw from the study at any time. However, if you do not want the researchers to use or disclose any further information in this study you must cancel permission in writing and may do so at any time. If you cancel your permission, you will stop taking part in the study and no new information will be collected about you. However, if you cancel your permission, it will not apply to actions already taken or information already collected about you by the hospital or the researchers before you canceled your permission.

Generally, the entire research record and any medical records held by the hospital may be used and released for research purposes. The following people or businesses/companies/ might use, release, or receive such information:

- The researcher and their support staff;
- The study sponsor, the Rhode Island Neuroscience Leadership Committee;
- Doctors, nurses, laboratories and others who provide services to you or the sponsor in connection with this study;
- The company or section of the U.S. government that is paying for the study and others they hire to oversee, administer, or conduct the research;
- The United States Food and Drug Administration, the Department of Health and Human Services, the Office of Inspector General, and the Office of Civil Rights; European Medicines Agency
- People who volunteer to be patient advocates or research volunteer protectors;
- Members of the hospital's administrative staff responsible for reviewing, approving and administering clinical trials and other healthcare or research activities.
- Accrediting Organizations

There are times when the law might require or permit Lifespan to release your child's health information without your permission. For example, Rhode Island law requires researchers and health care workers to report abuse or neglect of children to the Department of Children, Youth and Families (DCYF) and to report abuse or neglect of people age 60 and older to the Department of Elderly Affairs.

All researchers and health care providers are required to protect the privacy of your child's health care information. Other people and businesses/organizations that are not health care providers are not required by law to do that so it is possible they might re-release your child's information.

You have the right to refuse to sign this form and not allow your child to participate in the research. Your refusal would have no effect on your child's treatment, charges billed to you, or benefits at any Lifespan health care site. If you do not sign, your child will not be able to enroll in the research study and will not receive treatment as a study participant.

If you decide to have your child quit the study after signing this form (as described in Section 6) no new information will be collected about them unless you gave us permission to do so. However, the hospital or the researchers may continue to use information that was collected before you removed your child from the study to complete analysis and reports of this research.

For more detail about privacy rights see the Lifespan Joint Privacy Notice which has or will be given to you.

#### FUTURE RESEARCH

It is possible that your child may be eligible for another research study in the future. The researchers are requesting your permission to contact you to find out if you are interested in having your child participate in any future studies. Please place your initials next to one of the boxes below to tell the study team whether or not you want to be contacted about future research studies.

| | I DO want to be contacted about future studies. |
|------------|-----------------------------------------------------|
| (Initials) | _ |
| | I DO NOT want to be contacted about future studies. |
| (Initials) | |

## **SIGNATURE**

I HAVE READ THE ABOVE DESCRIPTION OF THIS STUDY. ALL OF MY QUESTIONS HAVE BEEN SATISFACTORILY ANSWERED, AND, AND I GIVE PERMISSION FOR MY CHILD TO PARTICIPATE IN THIS RESEARCH STUDY.

This informed consent document does not have an expiration date.

| The Researcher is required to provide a | copy of | this co | onsent to you. |
|---|---|---|---|
| Signature of parent/guardian* | Date | and | Time when signed |
| Signature of parent/guardian* | Date | and | Time when signed |
| I AGREE TO PARTICIPATE IN THIS STUDY | | | |
| Signature of study volunteer (child)* | Date | | |
| Age of study volunteer (child) | | | |
| I WAS PRESENT DURING THE CONSENT PR<br>AGREEMENT ABOVE BY THE PARENT/GUA<br>REPRESENTATIVE | | | |
| Signature of witness (required if consent presented orally or at the request of the IRB) | | Date | |
| Signature of Translator | | Date | |

| IF STUDY VOLUNTEER IS UNABLE TO SIGN OR EXCEPTION TO ASSENT IS SOUGHT, PLEASE EXPLAIN: |
|---|
| I CERTIFY THAT I HAVE EXPLAINED FULLY TO THE ABOVE PARENTS AND STUDY VOLUNTEER, THE NATURE AND PURPOSE, PROCEDURES AND THE POSSIBLE RISK AND POTENTIAL BENEFITS OF THIS RESEARCH STUDY. |
| Signature of researcher or designate Date and Time when signed |
| * If signed by agent other than parent and study volunteer, please explain below. |